CLINICAL TRIAL: NCT00148304
Title: Insulin Treatment Variation in Southwestern Diabetics - Therapeutic Decision-making
Brief Title: Insulin Treatment Variation in Southwestern Diabetics
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 04-176
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes; Self-Monitoring, Blood Glucose
Keywords: Decision-making; Insulin; Preference; Treatment Variation; Provider; Patient
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The purpose of this study is to better understand disparities in insulin dosing, hemoglobin A1c, and self-reported patient self-care behaviors among non-Hispanic white, Hispanic, and African American veterans with type 2 diabetes receiving VA care.

DETAILED DESCRIPTION:
Background: Minority populations are disproportionately affected by type 2 diabetes mellitus (T2DM), likely due to an interaction of genetic and environmental risk factors. Several studies have documented a higher prevalence of insulin resistance, disparities in quality of care, and more microvascular and macrovascular complications in minority groups. Recent evidence by our research group indicates that insulin-using minority veterans have poorer glycemic control (as measured by HbA1c) and receive lower doses of insulin than do non-Hispanic white patients.

Objectives: The goal of this mixed methods descriptive, cross-sectional study is to elucidate the patient, provider and interactive patient/provider reasons for this discrepancy, to determine and validate these findings in a much larger sample, and to use what is discovered to develop strategies to remedy provider and patient behaviors in order to optimize health outcomes. The objective of this mixed method study is to unpack provider decision-making and patient self-care behaviors responsible for ethnic and racial variation in the use of insulin in veterans with T2DM receiving VA care, while adjusting for important covariates and confounders. Aim 1: Perform a qualitative provider Nominal Group Technique designed to elucidate insulin prescribing decision-making behaviors, and possible reasons for racial/ethnic variation in insulin use. Aim 2: Perform a qualitative content analysis of patient focus group data on insulin-using veterans in VA care across African American, Hispanic and non-Hispanic White (NHW) contrasts. Psychosocial determinants of self-care, diabetes care preferences, patient/provider relationship issues, and possible reasons for racial/ethnic variation in insulin use will be explored. Aim 3: Construct a) patient, and b) provider questionnaires reflective of qualitative focus group data, nominal group process and extant evidence-base findings, and Aim 4: Administer surveys to a) a racially/ethnically diverse random sample of insulin-using diabetic veterans receiving care within VISN 18, and b) their assigned primary care providers.

Methods: This is a mixed methods descriptive, cross-sectional study using 1) qualitative nominal group technique data (from providers), focus group data (from patients) and 2) provider and nested patient survey data. The investigators will use qualitative methods to explicate and deconstruct the etiologic associations and management strategies of insulin-using patients and their providers using focus group content analytical methods. Next, the investigators will use the extant evidence from the evidence-base, focus group data and conventional survey methods to construct two surveys-one targeted to providers and another to survey a randomly selected population of representative veterans nested within their providers VA care, following the recommendations of Hughes, O'Brien and Dillman.

Status: Completed.

ELIGIBILITY:
Inclusion Criteria:

* Must be in VISN 18 VISTA database
* Diabetic
* Using insulin

Exclusion Criteria:

- Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: insulin-using diabetics in VISN 18
Sampling Method: Non-Probability Sample
Enrollment: 1248 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
diabetes self-care/attitudes | single survey

CONTACTS AND LOCATIONS:
Overall Officials: Glen H Murata, MD, Principal Investigator — New Mexico VA Health Care System, Albuquerque, NM
Locations (3):
- United States (3):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico